CLINICAL TRIAL: NCT03648749
Title: Evaluation of a Speech-to-noise Feedback Device for Treatment of Hypophonia in Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: University of Western Ontario, Canada (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LawsonHRI5264; 111861 (Other: Western University Health Sciences Research Ethics Board)
Record Dates: First submitted 2018-08-22; First posted 2018-08-27 (Actual); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: A single group will be studied during no intervention (no feedback about speech) and intervention (feedback about speech) phases.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Speech-to-noise feedback (Experimental): A target speech-to-noise level is specified and feedback about achievement of the target level is provided
  Interventions: Behavioral: Speech-to-noise feedback

INTERVENTIONS:
Behavioral: Speech-to-noise feedback — A target speech-to-noise level is specified and feedback about achievement of the target level is provided.

SUMMARY:
This study will evaluate the effectiveness of a speech-to-noise feedback procedure for the treatment of hypophonia in Parkinson's disease. The procedure includes a device that records the sound intensity level of the wearer's speech and compares it to the noise level around them. The device will provide the wearer with feedback if their speech becomes too quiet for them to be heard by their listener.

DETAILED DESCRIPTION:
This study will evaluate the effectiveness of a speech-to-noise feedback procedure for the treatment of hypophonia in Parkinson's disease. The procedure includes a device that records the sound intensity level of the wearer's speech and compares it to the noise level around them. The device will provide the wearer with feedback if their speech becomes too quiet for them to be heard by their listener.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with idiopathic Parkinson's disease and hypophonia by a neurologist at least 6 months prior to participation.
* stabilized on antiparkinsonian medication.
* good general health.
* pass a 40 decibel hearing screening.
* proficient enough in English to participate in speech testing.

Exclusion Criteria:

* history of stroke or an additional neurological or motor control disorder.
* history of speech impairment that is unrelated to Parkinson's disease.

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2019-03-01 (Estimated); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Average speech-to-noise ratio | Single two-hour visit.
  Average speech-to-noise ratio value will be obtained over a two-hour interval.

SECONDARY OUTCOMES:
Percent Speech Intelligibility Score (PSIS) | Single two-hour visit.
  PSIS is the percentage of words that can be correctly understood by a person listening (listener) to the participant's speech while they read sentences aloud. The PSIS ranges from 0% to 100%. This is a total score. Higher PSIS are considered better. The PSIS are obtained using communication partners (i.e. spouse) who listen and provide live repetitions of the spoken sentences. The spoken repetitions are transcribed by the investigators and compared to the printed reading material to calculate the percent of correctly transcribed words. The result is the PSIS referenced to a familiar listener (i.e. communication partner). The participant's spoken sentences are audio recorded and played to naïve listeners who provide written transcriptions of the participant's spoken sentences. The naïve listener transcribed sentences are compared to the printed reading material and the percent of correctly transcribed words is calculated. The result is the PSIS referenced to a naïve listener.
Ratings of Experience with the Device | Single two-hour visit.
  Participants rate their device experience with 5 visual-analogue scales (VAS) for 5 parameters. Participants see a 10cm horizontal line with end points and place a vertical line for their rating. Left is a poorer rating and right is a better rating. Parameter 1 is 'physical comfort' with left as 'uncomfortable' and right as 'comfortable'. Parameter 2 is 'visual presentation' with left as 'unacceptable' and right as 'acceptable'. Parameter 3 is 'response to feedback' with 'bothersome' (left) and 'not bothersome' (right). Parameter 4 is 'speech intensity' with 'too quiet' (left) and 'too loud' (right). Parameter 5 is 'overall preference' with 'low preference' (left) and 'high preference' (right). Vertical lines placed on the VAS are measured by hand from the left end and expressed as percent of the total VAS line. The 5 device experience parameter ratings are expressed as separate percentage VAS scores and will not be used to calculate a total score.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Adams, PhD, Principal Investigator — Western University
Locations (1):
- LawsonHRI, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No